CLINICAL TRIAL: NCT04043871
Title: Concordance Between the Foot-to-Apex Systolic Interval and the Auscultatory Method for Measurement of Brachial Systolic Pressure in Patients With Severe Renal Failure: Pilot Study
Brief Title: Concordance Between the Foot-to-Apex Systolic Interval and the Auscultatory Method for Measurement of Brachial Systolic Pressure in Patients With Severe Renal Failure
Acronym: SFATI-IRC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Technology Transfer Accelerator Offices _ SATT AxLR (Unknown)
Responsible Party: Sponsor
Other Study IDs: IDIL/2018/APM-02; 2018-A03347-48 (Other: ANSM)
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2019-05

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with renal insufficiency
  Interventions: Diagnostic Test: Systolic blood pressure

INTERVENTIONS:
Diagnostic Test: Systolic blood pressure — Systolic blood pressure measured by Foot-to-Apex Systolic Interval, conventional oscillometric measurement, and the auscultatory method

SUMMARY:
The investigators hypothesize that the Systolic Foot-to-Apex Time Interval (SFATI) method will be accurate for measurement of systolic blood pressure with marked arterial stiffness as seen in patients with severe renal impairment. Also that the presence of arterial calcifications only changes the agreement between the SFATI method and the reference method (auscultatory method) if the calcifications are very severe.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient under consultation in the Nephrology for severe renal impairment (defined by a glomerular filtration rate <30 mL / min, assessment within previous 3 months)

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with severe renal impairment (defined by a glomerular filtration rate <30 mL / min, assessment within previous 3 months), stage 4 or stage 5.
  Patients will be selected during consultations in the Nephrology department or during dialysis sessions at the University Hospital of Nîmes.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure according to oscillometric curve | Day 0
  mmHg measured by Systolic Foot-to-Apex Time Interval
Systolic blood pressure according to Korotkov sounds | Day 0
  mmHg measured by auscultatory method

SECONDARY OUTCOMES:
Brachial pulse wave velocity | Day 0
  m/s
Systolic blood pressure according to conventional oscillometric measurement | Day 0
  mmHg; Dinamap
Brachial artery calcium score | Day 0
  Measured by ultrasound of the arteries of the upper limb
Presence of arterial rigidity | Day 0
  Yes/No, measured by Complior > 10 m/s
Disease-associated patient characteristics | Day 0
  Age, sex, diabetes, Chronic Renal Disease stage
Modification of antihypertensive treatment to maintain systolic tension between 110 and 130 mm Hg | Day 0
  Change in antihypertensive treatment following measurement

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez Martin, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Result] Benmira AM, Moranne O, Prelipcean C, Pambrun E, Dauzat M, Demattei C, Perez-Martin A. Direct Determination rather than Oscillometric Estimation of Systolic Blood Pressure in Patients with Severe Chronic Kidney Disease. Am J Nephrol. 2022;53(1):41-49. doi: 10.1159/000520996. Epub 2022 Jan 12. PMID 35021175